CLINICAL TRIAL: NCT01994564
Title: Prevalence of Dyschromatopsia in Glaucoma Patients
Status: Withdrawn | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Other Study IDs: 356715-1 Dyschromatopsia
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2012-07

CONDITIONS: Open Angle Glaucoma
Keywords: OAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is a progressive disease resulting in loss of retinal nerve cells and their axons (retinal nerve fibers). Retinal nerve fibers are ordered in a special manner when they enter the optic nerve. Hence, damage to the retinal nerve fibers by glaucoma results in visual field defects at certain locations. Furthermore, the retinal nerve fiber layers from different receptors for different colors are ordered in a special manner as well. Thus, it is possible that glaucomatous damage causes color vision dysfunction (dyschromatopsia).

At the moment there is disagreement whether dyschromatopsia occurs at early- to mid-stage or only in end-stage glaucoma.

By testing color vision in glaucoma patients the prevalence of dyschromatopsia in glaucoma and in different stages of the disease will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of open angle glaucoma
* visual acuity >/= 20/50
* age >/= 18 (no upper limit)
* male or female gender

Exclusion Criteria:

* other type of glaucoma
* age <18
* other retinal disease (e.g. age related macular degeneration)
* other disease affecting the optic nerve or the retinal nerve fibers
* known color blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of open-angle glaucoma of the Glaucoma Department at Massachusetts Eye & Ear Infirmary, Boston, MA 02114, US
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Result from Ishihara Test | Visit 1
  Color vision will be tested once by Ishihara plates. Both eyes will be tested separately.

SECONDARY OUTCOMES:
Glaucoma stage | Visit 1
  Visual field will be tested with 30-2 Humphrey visual field full threshold test. Visual field defects will we graded following the Hodapp-Anderson-Parrish Scale (Hodapp E, Parrish RK, Anderson DR. Classification of Defects in Clinical Decisions in Glaucoma. St. Louis: Mosby, 1993:52-61).

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J. Rhee, M.D., Principal Investigator — Massachusetts Eye & Ear Infirmary, Harvard Medical School, Boston, MA, US
Locations (1):
- Massachusetts Eye & Ear Infirmary, Boston, Massachusetts, United States